CLINICAL TRIAL: NCT01811914
Title: Intraoperative Focused TTE - Impact on High Risk Patients´ Management in Hemodynamic Instabilities
Brief Title: Focused TTE for Hemodynamic Instable High Risk Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philipps University Marburg (Other)
Collaborators: Kerckhoff Heart Center (Other)
Responsible Party: Principal Investigator, Dr. Thomas Kratz, Dr. Thomas Kratz, Philipps University Marburg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UKGMTTE4
Record Dates: First submitted 2013-03-13; First posted 2013-03-15 (Estimated); Last update posted 2014-04-17 (Estimated); Status verified 2014-04

CONDITIONS: Hemodynamic Instability During Anesthesia; High Risk Surgery
Keywords: focused TTE; intraoperative TTE; transthoracic echocardiography; high risk non-cardiac surgery; hemodynamic instabilities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- intraoperative TTE (Experimental): TTE if a hemodynamic instability occurs
  Interventions: Other: intraoperative TTE

INTERVENTIONS:
Other: intraoperative TTE
  Other Names: focused transthoracic echocardiography; focused TTE; intraoperative transthoracic echocardiography

SUMMARY:
Focused transthoracic echocardiography (TTE) is a technique, which allows quick and non-invasive diagnosis and monitoring in hemodynamic instable patients. There are preliminary data supporting the hypothesis that TTE is feasible in the operating theatre.

The purpose of this study is to test the hypothesis that intraoperative focused TTE has an impact on high risk patients´ management when it is added to standard extended monitoring practices in hemodynamic instabilities.

DETAILED DESCRIPTION:
Focused TTE is en emerging matter in anesthesia, intensive care and emergency medicine. The value of intraoperative TTE is unclear. There are preliminary data that it is feasible For intraoperative transesophageal echocardiography (TEE) an impact on cardiac and non-cardiac surgery patients´ management has been shown.

Purpose of this study is to evaluate the application of focused TTE in patients with increased perioperative risk undergoing moderate to high risk surgery who become hemodynamic instable during anesthesia in the operating theatre.

When hemodynamic instability under anesthesia occurs focused TTE is conducted and the obtained diagnostic information are used for further patient management. Any change in management or therapy will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* gender: male, female
* Age ≥ 18 years
* increased perioperative risk, at least one of the following:

  * coronary artery disease
  * congestive heart disease
  * insulin dependent diabetes mellitus
  * renal insufficiency, creatinine > 2,0 mg/dl
  * cerebrovascular disease
  * Sepsis
* Procedure with at least moderate increased risk

  * intraperitoneal surgery
  * intrathoracal surgery
  * major orthopedic/traumatologic surgery
  * prostatic surgery
  * vascular surgery
* Hemodynamic instability, at least one of the following:

  * Hypotension (systolic blood pressure < 80 mmHg or mean blood pressure <50 mmHg) and/or
  * Bradycardia < 45/min. orr Tachycardia > 120/min and/or
  * Cardiac index < 2,0 l/min/m2

Exclusion Criteria:

* cardiac surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-03; Primary Completion 2013-11 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Change of patients´ management | at time of anesthesia / surgery
  Recordings of TTE findings influencing change of patient´s management in the operating theatre

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Kratz, MD, Principal Investigator — Department of Anesthesia and Intensive Care Medicine, University Hospital Marburg, Germany
Locations (1):
- University Hospital of Marburg, Department of Anesthesia, Marburg, Germany